CLINICAL TRIAL: NCT00323999
Title: A Randomised Trial to Compare the Differences Between Monopolar Surgery (Loop Resection) With Glycine 1,5% and Bipolar Surgery With Saline (Olympus,Versapoint) on Hysteroscopic Surgery.
Brief Title: Hysteroscopic Monopolar and Bipolar Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Other Study IDs: AB170262
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2006-05-10 (Estimated); Status verified 2006-05

CONDITIONS: Menorrhagia; Fibroid; Polyps
Keywords: Hysteroscopic resection; Menorrhagia; fibroids; polyps
MeSH Terms: conditions — Menorrhagia; Leiomyoma; Polyps | interventions — Endomet

INTERVENTIONS:
Procedure: Hysteroscopic resection of fibroids, polyps and endometrium.

SUMMARY:
The aim of the study is to evaluate bipolar equipment versus monopolar, and to see if there is any differences between the two types of bipolar equipment espescially regading both safety and effect.

DETAILED DESCRIPTION:
* Trial design: A prospective randomised study with three arms, one arm with monopolar surgery and two different arms with bipolar surgery. Its a one center study.
* Trial population: Pre-or perimenopausal women reffered to our clinic with bleeding disorders and were we plan to do endometrial resection. Patients with a bleeding disorder due to fibroids type 0 and 1 will be included and patients with polyps were endometrial resection is planned at the same time will also be included.
* Preoperative selection: The fibroids will be mapped using transvaginal ultrasound according to the classification ESGE. Type 0 and 1 fibroids will be included. Diameter of the fibroid must not extend 4cm. The endometrium size double layer will be recorded. Uterine size anetrior /posterior diameter, longitudinal diameter (cavity; top fundal to isthmus) will be measured. Were polyps are included these will be measured; length and width. Higham score (PBAC), Se-hgb, Ferritin, FSH and Oestradiol will be documented at all visits. Menstrual pain will be documented due to a VAS-scale.
* Treatment regimen:Randomisation in blocs of 20 between monopolar and two types of bipolar surgery.
* Surgical Technique: The cervical canal will be dilated to Hegar 10 or 11 and a rigid resectoscope Ch. 26 is passed to the uterine cavity. Glycine 1,5% or Saline (Baxter) is infused to irrigate the uterine cavity (Iglesias technique) Automatic pressure cuff maintains an infusion pressure of 100mm Hg and suction 10-15mmHg is applied to the outflow tube in order to achieve a sufficient flow.Fibroids type 0 and 1 are resected in total if possible or flush to the plane of the uterine wall. The tissue chips are removed at intervals by currette and forceps. The operation will be performed by experienced surgeons.
* Primary response variables: Safety is our primary response variable. Fluid absorption and lowering of Se-Sodium will be analysed. These parameters are the only objective parameters which can tell us about safety. Nausea will be reorded on a VAS-scale.

  * Secondary resonse variables: Operating time, tissue removed, easisness of operation, levels of vaginal bleeding measured by the methosd of Hgham(PBAC)before and at follow up.

After 6 month and one year we will look at secondary intervention like repeated resection or hysterectomy.

ELIGIBILITY:
Inclusion Criteria:-Pre-or perimenopausal women with a bleeding disorder with or without fibroids or polyps -

Exclusion Criteria:-Postmenopausal patient. Infertility. Additional condition requiring treatment detected during examination. Malignancy or atypical hyperplasia detected by histological examination.

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2004-12; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Olav Istre, MD., PhD., Principal Investigator — Department of Gynaecology, Ullevaal University Hospital, Oslo, Norway
Locations (1):
- Gynaecological department Ullevaal University Hospital, Oslo, Norway